CLINICAL TRIAL: NCT04931433
Title: Intravenous Lignocaine as an Analgesic Adjunct in Adolescent Idiopathic Scoliosis Surgery (IGNITE-AIS Study)
Brief Title: Intravenous Lignocaine as an Analgesic Adjunct in Adolescent Idiopathic Scoliosis Surgery
Acronym: IGNITE-AIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UM.M/PDR/638/3(151)
Record Dates: First submitted 2021-01-24; First posted 2021-06-18 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Adolescent Idiopathic Scoliosis; Analgesia
Keywords: Intravenous Lignocaine; Post-operative pain; Posterior Spinal Fusion; Pharmacokinetics
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Group A, Lignocaine and Group B, placebo. Group A will receive 1.5 mg/kg IV lignocaine bolus prior to induction followed by 2mg/kg/hour of lignocaine infusion throughout surgery until wound closure in which the infusion rate will be halved to 1 mg/kg/hour until the end of surgery. This same rate will be infused in the recovery room for another half an hour before patient discharge. Group B will receive saline of similar volume and rate as for Group A.
Who Masked: Participant, Outcomes Assessor
Masking Description: The medications will be prepared before induction by a nurse or doctor who is neither a member of the trial team and later handed to the anaesthetist in charge of the administration according to the trial protocol. The trial drugs are prepared in a 10-ml syringe for the bolus injection and a 50-ml syringe for continuous infusion. For the bolus injection, IV lignocaine 1% will be drawn into the 10-ml syringe will lignocaine 1% solution according to the weight of the patient (0.15ml/kg) or an equal amount of 0.9% saline. The 50-ml syringe contained either 50ml of lignocaine 1% solution or 0.9% normal saline solution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lignocaine (Experimental): This arm will receive intravenous Lignocaine bolus and infusion
  Interventions: Drug: Lignocaine
- Placebo (Placebo Comparator): This arm will receive Normal saline 0.9% bolus and infusion
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lignocaine — Group A will receive 1.5mg/kg IV lignocaine bolus prior to induction followed by 2mg/kg/hour of lignocaine infusion throughout surgery until wound closure in which the infusion will be halved to 1mg/kg/hour until the end of surgery. The same rate will be infused in the recovery room for another half an hour before participant is discharge.
  Other Names: Group A
  Arms: Lignocaine
Drug: Normal saline — Group B will receive saline of similar volume and rate as Group A
  Other Names: Group B
  Arms: Placebo

SUMMARY:
This is a single-center study comparing the effect of intravenous (IV) Lignocaine given throughout posterior spinal fusion surgery on the reduction of morphine usage during postoperative period in adolescent idiopathic scoliosis (AIS) patients.

DETAILED DESCRIPTION:
Study Rationale

Posterior spinal fusion (PSF) performed for the correction of adolescent idiopathic scoliosis (AIS) is a complex surgery which result in severe postoperative pain. Early and adequate analgesia facilitates early mobilization hence reduces postoperative complications. Multimodal analgesia technique has been shown to improve perioperative pain management and significantly reduced the opioid usage and its side effects. Intravenous lignocaine infusion has been used as an analgesic adjunct for the management of acute postoperative pain in many clinical settings which include adult complex spinal surgery. However, until this date no study which examines AIS patients undergoing PSF surgeries.

Study Design

This is a prospective, double-blinded, randomized placebo-controlled trial. Participants will be randomized using a sequentially numbered, opaque sealed envelope (SNOSE) method into two groups: Group A, Lignocaine and Group B, placebo. Group A will receive 1.5mg/kg IV lignocaine bolus prior to induction followed by 2mg/kg/hour of lignocaine infusion throughout surgery until wound closure in which the infusion rate will be halved to 1mg/kg/hour until the end of surgery. The same rate will be infused in the recovery room for another half an hour before patient discharge. Group B will receive saline of similar volume and rate as for Group A.

Study Intervention

The trial drugs are prepared in a 10-ml syringe for the bolus injection and an 50-ml syringe for continuous infusion. For the bolus injection, IV lignocaine 1% will be drawn into the 10-ml syringe according to the weight of the patient (0.15ml/kg) or an equal amount of 0.9% saline. The 50-ml syringe will contained either 50ml of lignocaine 1% solution or 0.9% normal saline solution. Both syringes will be labeled as Drug X.

The depth of anesthesia will be monitored using a processed electroencephalogram (EEG) monitor called Conox (commercial brand name of Fresenius Kabi, Germany depth of anesthesia monitor). There are two indices, the qCON which is the index of hypnotic effect and the qNOX which is the index of pain/nociception. A qCON value of 40-60 indicates general anesthesia state and a qNOX value of 40-60 implies that patient is unlikely to respond to noxious stimuli.

Continuous monitoring of patients will be carried out using invasive blood pressure via radial artery cannulation, heart rate, pulse oximetry and 3-lead electrocardiogram. All participants will be operated utilizing a dual attending surgeon strategy involving two senior surgeons. Intraoperative neurophysiological monitoring using somatosensory and motor evoked potentials will be used throughout the surgery.

All patients will be adequately fasted for at least 6 hours prior to surgery without premedication. The trial drug will be administered to the participants according to the allocation. The bolus injection will be administered over 3 minutes prior to induction followed by an infusion as per protocol. Induction of anesthesia will be performed with IV Target Controlled Infusion (TCI) of Propofol 4-6mcg/ml and TCI Remifentanil 3-5ng/ml. After tracheal intubation, patients will be ventilated with 50% Oxygen/air mixture and anesthesia is maintained with TCI Propofol 2-4mcg/ml and TCI Remifentanil 2-5ng/ml. A qCON value of 40-60 will be targeted intraoperatively. IV Dexamethasone 4mg and IV Morphine 0.5mg/kg will be administered prior to skin incision.

During the maintenance phase of anesthesia if the qCON value is outside this range for longer than 10 seconds, the concentration of Propofol will be increased or decreased by 0.5mcg/ml. After the new target concentration is reached, an additional 20 seconds will be given to bring the qCON value within the pre-established range before making further adjustments.

Upon wound closure, additional IV Morphine 0.5mg/kg will be administered with IV acetaminophen 15mg/kg and IV Ondansetron 0.15mg/kg. IV Fentanyl 0.5mcg/kg will be given prior to cessation of TCI Remifentanil at skin closure. TCI Propofol will be ceased once skin closure is completed. Participants are extubated in the operation room after completion of surgery and transfer to recovery bay for monitoring. The time of discontinuation of TCI Propofol (T0) and the time elapsed from T0 to extubation will be recorded. The qCON value at extubation will be recorded.

The trial drug is continued up to 30 minutes post-operation in the recovery room. Sedation score will be assessed using Richmond Analgesia Sedation Scale (RASS) at the interval of 15 minutes. Pain score will be evaluated using Numerical Rating Scale (NRS) at the interval of 10 minutes. Rescue bolus of IV Fentanyl 10mcg will be given every 5 minutes to treat breakthrough pain when pain score is >=4. Once the pain score is <4, Patient Controlled Analgesia (PCA) with morphine will be started at a concentration of 2mg/ml, a demand dose of 1mg/ml with a lockout interval of 5 minutes and a maximum dose of 20mg over 4 hours without background infusion.

Postoperative analgesia will be maintained using multimodal strategy. Participants will be continued on PCA morphine for up to 48 hours. Participants will receive IV acetaminophen 15mg/kg every 6 hours for the first 24 hour and changed to oral thereafter and oral Celebrex 200mg daily (for <35kg) or 200mg every 12 hours (for >= 35kg), NRS will be recorded every 4 hours until the patient is discharged.

Measurement of Plasma Concentration Levels of Lignocaine

5mls of blood samples will be collected from participants using Ethylenediaminetetraacetic acid (EDTA) tube 30 minutes, 2 hours, 4 hours and 8 hours after the bolus injection. Collected blood samples will be centrifuged immediately and the plasma will be transferred into cryo vials in duplicates and kept at -80 degree Celsius until further analysis.

To extract lignocaine from plasma 0.5ml volume of plasma, 0.1ml internal standard (IS) solution (500ng/ml), 0.1ml 1Molar of Sodium Hydroxide (NaOH) and 3ml of methyl-tert-butyl ether (MTBE) will be placed in a 4.5ml propylene tube. The content will be mixed for the minimum of 5 minutes by the shaker and then centrifuged at 3000-3500rpm for 5 minutes. The top layer will be transferred to a 4.5ml propylene tube containing 0.25ml of 0.1% Formic acid. The tube will be mixed again for the minimum of 5 minutes by the shaker and then centrifuge at 3000-3500rpm for 5 minutes. The top solvent layer will be discarded by vacuum and the remaining solution will be transferred into an autosampler vial. A 100 microliter volume will be injected into the analytical column connected to light chain mass spectrometry system. The calibration curve will be plotted by the ratio of the lignocaine/IS vs the concentration of lignocaine. The concentration of lignocaine in all samples will be calculated from the calibration curve.

Data Analysis

All data will be tabulated in a computer files and analyzed using International Business Machines Statistical Package for the Social Sciences (IBM SPSS) software version 25. All randomized participants will be analyzed according to their original allocation according to the (modified) intention-to-treat principle except those who deemed ineligible after randomization or the treatment is never started (such as last minute cancellation of surgery). Data normality will be assessed by using the Kolmogorov-Smirnov test and confirm with visual inspection of the histogram. Categorical data will be presented as counts and percentage. Continuous date will be expressed as mean +/- standard deviation, or median (Q1-Q3) for data with skewed distribution. Data differences between the two groups will be computed by independent t-test or Mann Whitney U test for continuous data and the Chi square test for categorical data.

The mean plasma concentration of lignocaine will be plotted against time from bolus injection and during continuous infusion perioperatively until the infusion is discontinued.

The primary outcome, postoperative morphine consumption at 24 hour and Propofol requirements between group, will be analyzed by using independent t-test. Mixed analysis of variance (ANOVA) will also be conducted to determine whether the change in the use of PCA morphine over time (at 12 hours, 24 hours, 36 hours and 48 hours post-surgery), the change in target effect site concentration of Propofol and remifentanil and qCON value over time are the result of the interaction between the two groups and time. If an interaction is present, the differences between group at each time point will be calculated and compared by using the independent t-test; however, if no statistical interaction is present, the main effects of the analysis will be reported. The occurrence of adverse events or complications will be compared between group by using the Chi square test. A Kaplan-Meier analysis will be conducted for time-to-first flatus, time-to-first ambulation and time to recovery from anesthesia and will be compared between group using Mantel-Cox test. A 2-sided p<0.05 is considered statistical significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status I and II

Exclusion Criteria:

* Hypersensitivity to amide local anaesthetics/lignocaine
* Liver disease (alanine aminotransferase, ALT or aspartate aminotransferase, AST more than twice normal)
* Renal impairment (defined as estimated Glomerular Filtration Rate <= 60ml/min)
* History of cardiac disease/cardiac arrhythmia
* Epilepsy
* Intellectual disability
* Preoperative chronic pain with regular opioid usage

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
To evaluate postoperative morphine consumption at 24 hours | Immediately post-operation until 24 hours post-operation
  Amount of patient controlled analgesia (PCA) morphine usage in mg over 24 hours

SECONDARY OUTCOMES:
To determine the safe dose of intravenous infusion (IVI) lignocaine by measuring the plasma concentration levels | 30 minutes, 2 hours, 4 hours and 8 hours after the bolus dose of trial drug
  Blood sample either arterial (intra-operative) or venous (post-operative) will be collected and the plasma will be evaluated using Light Chain Mass Spectrometry to determine the concentration of lignocaine in the blood at specific time point
To evaluate the effect on propofol dose requirement as measured by processed electroencephalogram (EEG) qCON index | From the start of anaesthesia until the end of surgery (Throughout the surgery which may range from 2 to 5 hours))
  Total amount of propofol usage in milligram or the dose of propofol required throughout the surgery to maintain qCON value between 40-60 throughout the surgery will be documented and compared between 2 groups as lignocaine has been shown to have anaesthetic sparing effect. Processed EEG is an automated device of summation of raw EEG that generate dimensionless index value between 0 to 100. It does not specifically focus on single EEG waveform.

OTHER OUTCOMES:
To evaluate the postoperative numeric rating scale (NRS) at rest and during movement | Immediately after the operation until 48 hours after the operation
  Charting of numeric rating scale (NRS) at rest and during movement every 10 minutes at recovery room and 4 hourly in the ward will be compared between to 2 groups to evaluate the effectiveness of lignocaine as analgesic adjunct. The scale has a scale of 0 to 10. 0 is equivalent to no pain and scale of 10 is equivalent to severe and worst pain.
To determine any adverse events or complications following administration of systemic lignocaine until hospital discharge | The adverse event will be observed from the time of administration of study drug until the participants are discharge from hospital after the operation. (through the perioperative period, an average of 4 days)
  The incidence of any adverse event that occur including postoperative nausea and vomiting, perioral numbness and seizure, constipation will be recorded for all participants
To determine the effect of intravenous infusion (IVI) Lignocaine on postoperative return of bowel function | The observation will be done by calculating the hours after the surgery (from the start of postoperative time) to the return of passing first flatus as a measure of bowel opening, assessed up to 72 hours, whichever comes first
  We are comparing the rate of postoperative delay in returning of bowel habit between this two groups by measuring the time of participant passing first flatus after the surgery
To determine the effect of intravenous infusion (IVI) lignocaine on postoperative ambulation | The hours after the surgery (from the start of postoperative time) until the participants have their first ambulation will be calculated, assessed up to 72 hours, whichever comes first
  We are comparing the rate of postoperative delay in returning to normal activity specifically mobility in spine surgery as a consequences of inadequate pain control between the 2 groups by measuring the time of first ambulation for all participant
To evaluate the length of hospital stay | The number of days through hospital stay after the surgery (number of postoperative day in hospital), an average of 4 days
  To evaluate the impact of lignocaine as analgesic adjunct in the change of the number of days spent in the hospital for recovery after surgery
To evaluate the effect of lignocaine on intraoperative somatosensory evoked potential and motor evoked potential reading | The time starts from beginning of the surgery until the end of surgery (up to 300 minutes)
  To evaluate the effect of intravenous infusion (IVI) Lignocaine on the amplitude of both somatosensory and motor evoked potential reading recorded throughout the surgery and to compare the difference with placebo
To determine the hypnotic effect of lignocaine on recovery time from anaesthesia | The time starts from the discontinuation of TCI Propofol to the time participant is extubated from the endotracheal tube which may vary from 15 to 30 minutes
  Comparison will be made between both groups whether there is a delay in recovery from anaesthesia by recording the time taken (in minutes) for each participant to be fully awake and extubated from the endotracheal tube once the TCI Propofol is discontinued.
To determine the antinociceptive property of lignocaine as measured by qNOX value | The time starts from beginning of the surgery until the end of surgery (up to 300 minutes)
  qNOX value will be blinded throughout the surgery and will be separately recorded. The trend of this value will be compared between 2 groups whether lignocaine has significant effect on to lower the qNOX value

CONTACTS AND LOCATIONS:
Overall Officials: Mohd Shahnaz Hasan, Postgraduate, Principal Investigator — University of Malaya
Locations (1):
- University Malaya, Pantai Valley, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beilin B, Shavit Y, Trabekin E, Mordashev B, Mayburd E, Zeidel A, Bessler H. The effects of postoperative pain management on immune response to surgery. Anesth Analg. 2003 Sep;97(3):822-827. doi: 10.1213/01.ANE.0000078586.82810.3B. PMID 12933409
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Ben-Shlomo I, Tverskoy M, Fleyshman G, Cherniavsky G. Hypnotic effect of i.v. propofol is enhanced by i.m. administration of either lignocaine or bupivacaine. Br J Anaesth. 1997 Apr;78(4):375-7. doi: 10.1093/bja/78.4.375. PMID 9135355
- [Background] Himes RS Jr, DiFazio CA, Burney RG. Effects of lidocaine on the anesthetic requirements for nitrous oxide and halothane. Anesthesiology. 1977 Nov;47(5):437-40. doi: 10.1097/00000542-197711000-00010. PMID 911052
- [Background] Rehberg B, Xiao YH, Duch DS. Central nervous system sodium channels are significantly suppressed at clinical concentrations of volatile anesthetics. Anesthesiology. 1996 May;84(5):1223-33; discussion 27A. doi: 10.1097/00000542-199605000-00025. PMID 8624017
- [Background] Kim WY, Lee YS, Ok SJ, Chang MS, Kim JH, Park YC, Lim HJ. Lidocaine does not prevent bispectral index increases in response to endotracheal intubation. Anesth Analg. 2006 Jan;102(1):156-9. doi: 10.1213/01.ANE.0000184040.85956.98. PMID 16368822
- [Background] Myles PS, Leslie K, McNeil J, Forbes A, Chan MT. Bispectral index monitoring to prevent awareness during anaesthesia: the B-Aware randomised controlled trial. Lancet. 2004 May 29;363(9423):1757-63. doi: 10.1016/S0140-6736(04)16300-9. PMID 15172773
- [Background] Pandit JJ, Andrade J, Bogod DG, Hitchman JM, Jonker WR, Lucas N, Mackay JH, Nimmo AF, O'Connor K, O'Sullivan EP, Paul RG, Palmer JH, Plaat F, Radcliffe JJ, Sury MR, Torevell HE, Wang M, Hainsworth J, Cook TM; Royal College of Anaesthetists; Association of Anaesthetists of Great Britain and Ireland. 5th National Audit Project (NAP5) on accidental awareness during general anaesthesia: summary of main findings and risk factors. Br J Anaesth. 2014 Oct;113(4):549-59. doi: 10.1093/bja/aeu313. Epub 2014 Sep 9. PMID 25204697
- [Background] Hadley MN, Shank CD, Rozzelle CJ, Walters BC. Guidelines for the Use of Electrophysiological Monitoring for Surgery of the Human Spinal Column and Spinal Cord. Neurosurgery. 2017 Nov 1;81(5):713-732. doi: 10.1093/neuros/nyx466. No abstract available. PMID 29029325
- [Background] Haghighi SS, Madsen R, Green KD, Oro JJ, Kracke GR. Suppression of motor evoked potentials by inhalation anesthetics. J Neurosurg Anesthesiol. 1990 Jun;2(2):73-8. doi: 10.1097/00008506-199006000-00003. PMID 15815324
- [Background] Huotari AM, Koskinen M, Suominen K, Alahuhta S, Remes R, Hartikainen KM, Jantti V. Evoked EEG patterns during burst suppression with propofol. Br J Anaesth. 2004 Jan;92(1):18-24. doi: 10.1093/bja/aeh022. PMID 14665548
- [Background] Oliveira CM, Sakata RK, Slullitel A, Salomao R, Lanchote VL, Issy AM. [Effect of intraoperative intravenous lidocaine on pain and plasma interleukin-6 in patients undergoing hysterectomy]. Rev Bras Anestesiol. 2015 Mar-Apr;65(2):92-8. doi: 10.1016/j.bjan.2013.07.017. Epub 2014 Nov 7. Portuguese. PMID 25740274
- [Background] Kurabe M, Furue H, Kohno T. Intravenous administration of lidocaine directly acts on spinal dorsal horn and produces analgesic effect: An in vivo patch-clamp analysis. Sci Rep. 2016 May 18;6:26253. doi: 10.1038/srep26253. PMID 27188335
- [Background] Kandil E, Melikman E, Adinoff B. Lidocaine Infusion: A Promising Therapeutic Approach for Chronic Pain. J Anesth Clin Res. 2017 Jan;8(1):697. doi: 10.4172/2155-6148.1000697. Epub 2017 Jan 11. PMID 28239510
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Chan CYW, Kwan MK. Perioperative Outcome in Posterior Spinal Fusion for Adolescent Idiopathic Scoliosis: A Prospective Study Comparing Single Versus Two Attending Surgeons Strategy. Spine (Phila Pa 1976). 2016 Jun;41(11):E694-E699. doi: 10.1097/BRS.0000000000001349. PMID 26656053
- [Background] Kwan MK, Chan CY. Does a dual attending surgeon strategy confer additional benefit for posterior selective thoracic fusion in Lenke 1 and 2 adolescent idiopathic scoliosis (AIS)? A prospective propensity matching score analysis. Spine J. 2017 Feb;17(2):224-229. doi: 10.1016/j.spinee.2016.09.005. Epub 2016 Sep 5. PMID 27609611
- [Background] Miyabe M, Kakiuchi Y, Kihara S, Takahashi S, Kohda Y, Sato S, Toyooka H. The plasma concentration of lidocaine's principal metabolite increases during continuous epidural anesthesia in infants and children. Anesth Analg. 1998 Nov;87(5):1056-7. doi: 10.1097/00000539-199811000-00016. No abstract available. PMID 9806683
- [Result] Farag E, Ghobrial M, Sessler DI, Dalton JE, Liu J, Lee JH, Zaky S, Benzel E, Bingaman W, Kurz A. Effect of perioperative intravenous lidocaine administration on pain, opioid consumption, and quality of life after complex spine surgery. Anesthesiology. 2013 Oct;119(4):932-40. doi: 10.1097/ALN.0b013e318297d4a5. PMID 23681143
- [Result] Grassi P, Bregant GM, Crisman M. Systemic intravenous lidocaine for perioperative pain management: a call for changing indications in the package sheet. Heart Lung Vessel. 2014;6(2):137-8. No abstract available. PMID 25024999
- [Result] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Result] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Result] Greenwood E, Nimmo S, Paterson H, Homer N, Foo I. Intravenous lidocaine infusion as a component of multimodal analgesia for colorectal surgery-measurement of plasma levels. Perioper Med (Lond). 2019 Feb 26;8:1. doi: 10.1186/s13741-019-0112-4. eCollection 2019. PMID 30858969
- [Result] Both CP, Thomas J, Buhler PK, Schmitz A, Weiss M, Piegeler T. Factors associated with intravenous lidocaine in pediatric patients undergoing laparoscopic appendectomy - a retrospective, single-centre experience. BMC Anesthesiol. 2018 Jul 18;18(1):88. doi: 10.1186/s12871-018-0545-1. PMID 30021507
- [Result] Choi SJ, Kim MH, Jeong HY, Lee JJ. Effect of intraoperative lidocaine on anesthetic consumption, and bowel function, pain intensity, analgesic consumption and hospital stay after breast surgery. Korean J Anesthesiol. 2012 May;62(5):429-34. doi: 10.4097/kjae.2012.62.5.429. Epub 2012 May 24. PMID 22679539
- [Result] Bazin P, Padley J, Ho M, Stevens J, Ben-Menachem E. The effect of intravenous lidocaine infusion on bispectral index during major abdominal surgery. J Clin Monit Comput. 2018 Jun;32(3):533-539. doi: 10.1007/s10877-017-0035-x. Epub 2017 Jun 16. PMID 28623471
- [Result] Altermatt FR, Bugedo DA, Delfino AE, Solari S, Guerra I, Munoz HR, Cortinez LI. Evaluation of the effect of intravenous lidocaine on propofol requirements during total intravenous anaesthesia as measured by bispectral index. Br J Anaesth. 2012 Jun;108(6):979-83. doi: 10.1093/bja/aes097. Epub 2012 Apr 6. PMID 22490315
- [Result] Weber U, Krammel M, Linke S, Hamp T, Stimpfl T, Reiter B, Plochl W. Intravenous lidocaine increases the depth of anaesthesia of propofol for skin incision--a randomised controlled trial. Acta Anaesthesiol Scand. 2015 Mar;59(3):310-8. doi: 10.1111/aas.12462. Epub 2015 Jan 13. PMID 25582611
- [Result] Cui W, Li Y, Li S, Wang R, Li J. Systemic administration of lidocaine reduces morphine requirements and postoperative pain of patients undergoing thoracic surgery after propofol-remifentanil-based anaesthesia. Eur J Anaesthesiol. 2010 Jan;27(1):41-6. doi: 10.1097/EJA.0b013e32832d5426. PMID 19478674
- [Result] Hans GA, Lauwick SM, Kaba A, Bonhomme V, Struys MM, Hans PC, Lamy ML, Joris JL. Intravenous lidocaine infusion reduces bispectral index-guided requirements of propofol only during surgical stimulation. Br J Anaesth. 2010 Oct;105(4):471-9. doi: 10.1093/bja/aeq189. Epub 2010 Jul 21. PMID 20650919
- [Result] Senturk M, Pembeci K, Menda F, Ozkan T, Gucyetmez B, Tugrul M, Camci E, Akpir K. Effects of intramuscular administration of lidocaine or bupivacaine on induction and maintenance doses of propofol evaluated by bispectral index. Br J Anaesth. 2002 Dec;89(6):849-52. doi: 10.1093/bja/aef287. PMID 12453928
- [Result] Chen Z. The effects of isoflurane and propofol on intraoperative neurophysiological monitoring during spinal surgery. J Clin Monit Comput. 2004 Aug;18(4):303-8. doi: 10.1007/s10877-005-5097-5. PMID 15779842
- [Result] Urban MK, Fields K, Donegan SW, Beathe JC, Pinter DW, Boachie-Adjei O, Emerson RG. A randomized crossover study of the effects of lidocaine on motor- and sensory-evoked potentials during spinal surgery. Spine J. 2017 Dec;17(12):1889-1896. doi: 10.1016/j.spinee.2017.06.024. Epub 2017 Jun 27. PMID 28666848
- [Result] Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Weibel S. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Database Syst Rev. 2015 Jul 16;(7):CD009642. doi: 10.1002/14651858.CD009642.pub2. PMID 26184397
- [Result] Ibrahim A, Aly M, Farrag W. Effect of intravenous lidocaine infusion on long-term postoperative pain after spinal fusion surgery. Medicine (Baltimore). 2018 Mar;97(13):e0229. doi: 10.1097/MD.0000000000010229. PMID 29595671
- [Result] Maheshwari K, Avitsian R, Sessler DI, Makarova N, Tanios M, Raza S, Traul D, Rajan S, Manlapaz M, Machado S, Krishnaney A, Machado A, Rosenquist R, Kurz A. Multimodal Analgesic Regimen for Spine Surgery: A Randomized Placebo-controlled Trial. Anesthesiology. 2020 May;132(5):992-1002. doi: 10.1097/ALN.0000000000003143. PMID 32235144
- See also: Depth of anaesthesia monitors - Bispectral Index (BIS), E-Entropy and Narcotrend-Compact M — http://nice.org.uk/guidance/dg6